CLINICAL TRIAL: NCT07111091
Title: Comparison of the Effects of Unilateral and Bilateral Plastic Ankle Foot Orthosis on Gait and Balance in Children With Hemiparatic Cerebral Palsy
Brief Title: Effect of Ankle-Foot Orthosis on Gait and Balance in Children With Hemiparatic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yılmaz, Istanbul Medipol University, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 10840098604.01.01-E.56252
Record Dates: First submitted 2025-06-03; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy (CP); Hemiparatic Cerebral Palsy; Balance; Gait Analysis; Ankle Foot Orthosis (AFO)
MeSH Terms: conditions — Cerebral Palsy | interventions — Gait

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP A (Other)
  Interventions: Other: GAIT AND BALANCE EVALUATION
- GROUP B (Other)
  Interventions: Other: GAIT AND BALANCE EVALUATION

INTERVENTIONS:
Other: GAIT AND BALANCE EVALUATION — In our study, participants' walking assessments were made with GAITRite electronic walking path (CIR System INC. Clifton. NJ. USA.).
  In the postural balance assessments of the participants, the Bertec Balance Check Screener™ BP5050 20x20 inch (Bertec Comporation Columbus, OH, USA) force platform was used. The Bertec force platform is a three-component balance platform that is based on objectively measuring instantaneous changes in vertical force and center of pressure (CoP). Bertec was designed to evaluate the ability to maintain balance while standing.
  The assessments were made in all participants without an orthosis, with unilateral AFO and with bilateral AFO. In our study, participants were given a 10-minute rest period between assessments.

SUMMARY:
Background: Ankle-foot orthoses are frequently prescribed to reduce spasticity, position the extremity more properly, and regulate gait during the rehabilitation process of children with cerebral palsy.

Objective: To investigate the effects of unilateral or bilateral use of plastic ankle-foot orthoses (AFO) used in children with hemiparetic cerebral palsy (CP) on the child's gait and balance.

The aim of this study is to investigate the effects of unilateral and bilateral use of AFOs used in children with hemiparetic cerebral palsy on gait and balance.

Methods: 19 cooperative children aged 4-12 years, with gross motor function classification system levels 1 and 2, using bilateral AFOs were included in the study. Children were evaluated with bilateral AFOs, unilateral AFOs, and without AFOs. Trunk sway assessment was performed on the Bertec Balance force platform with eyes open and closed, and time-spatial characteristics of gait were evaluated with the GAITRite electronic walkway.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hemiparatic SP
* Cooperative
* Classified as 1 or 2 levels in GMFCS
* Lower extremity muscles with spasticity severity of up to 2 according to Modified Ashworth
* Using Bilateral Plastic AFO Orthosis for the last 6 months

Exclusion Criteria:

* foot deformity
* using walking aids
* unable to walk independently

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
balance | From enrollment to the end of treatment at 4 weeks
  Balance assessments were conducted using the Bertec Balance Check Screener™ force platform. Oscillations during the assessment were recorded for each participant. For safety reasons, the researcher stood close to the participant without contact during the balance assessment.

SECONDARY OUTCOMES:
demographic information form | From enrollment to the end of treatment at 4 weeks
  Orthosis information, including participants' full name, age, gender, weight, height, affected side, lower extremity length, and duration of orthosis use, was recorded.
Gait assessments | From enrollment to the end of treatment at 4 weeks
  In our study, participants' gait assessments were conducted using a GAITRite electronic walking path. Participants walked at a self-selected speed on a stable surface, while time and distance characteristics were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No